CLINICAL TRIAL: NCT00756587
Title: Cup Versus Bottle Feeding for Hospitalized Late Preterm Infants in Egypt
Brief Title: Cup Versus Bottle Feeding for Late Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Amel Abouelfettoh, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2004
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-09

CONDITIONS: Breastfeeding
Keywords: Cup Feeding; late Preterm
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Group one received feeding by bottle as the standard method of feeding in the NICU
  Interventions: Device: Bottle Feeding
- II (Experimental): Group 2 received all feeding by cup
  Interventions: Device: Cup Feeding

INTERVENTIONS:
Device: Cup Feeding — using a cup feeding technique for feeding the preterm infants during NICU stay
  Other Names: Cup-feeding Group
  Arms: II
Device: Bottle Feeding — receiving all feeding by bottle
  Other Names: bottle feeding group
  Arms: I

SUMMARY:
The purpose of the current study is to investigate the effect of using cup feeding for preterm infants during NICU stay on breastfeeding outcomes after discharge. The following hypotheses are being tested:

1. Infants Fed by cup during NICU stay will have higher breastfeeding proportions than infants fed by bottle
2. Infants fed by cup during NICU stay will have higher breastfeeding behaviour score on the Preterm Infant Breastfeeding Behavior Scale than infants fed by bottle

DETAILED DESCRIPTION:
The provision of breast milk is essential for preterm infants as it provides unique health benefits that are unmatched by other types of feeding [1-3]. However, breastfeeding presents unique challenges for preterm infants that include establishing and maintaining the mothers' milk supply and transitioning the infant from gavage feeding to breastfeeding [4]. One of the issues that presents during the transition to breastfeeding is that mothers of preterm infants are rarely available for all oral feedings during hospitalization; this makes it necessary for infants to receive oral feedings by other method, usually bottle feeding.

However, exposure of newborn infants to artificial nipples has been strongly associated with breastfeeding problems [5-9]. Frequently these problems have been explained by phenomena called nipple confusion. Nipple confusion occurs when infants are exposed to two different feeding methods, bottle and breast, resulting in the infant refusing to breastfeed. Consequently, it has been recommended that bottle feeding be avoided and that cup feeding be used for the supplementation of term as well as preterm infants.

Cup feeding is known as an alternative method of feeding breast milk to an infant using a small cup without a lip. Cup feeding is also recommended by the Baby Friendly Hospital Initiative.The use of cup was originally based on the goal of avoiding propping of bottles and also to increase bodily contact with the mother during feeding. Although cup feeding receives little mention in medical literature, and may seem to be a new technique for some, it has been used in several developing as well as developed countries. Lang, who observed cup feeding in South Nepal, implemented cup feeding in England and the practice expanded to other developed countries. Consequently cup feeding was established as a method for feeding infants who could not be breastfed from birth.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* 34 to 37 weeks of gestation at birth
* Maternal intention to breastfeed
* Fed only by tube feeding

Exclusion Criteria:

* Infants who had any condition interfering with oral feeding
* Infants with craniofacial anomalies
* Infants with intracranial hemorrhage

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2003-12; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Proportion | one week

CONTACTS AND LOCATIONS:
Overall Officials: Amel M Abouelfettoh, PhD, RN, Principal Investigator — Cairo University
Locations (1):
- Peiatric University NICU, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Abouelfettoh AM, Dowling DA, Dabash SA, Elguindy SR, Seoud IA. Cup versus bottle feeding for hospitalized late preterm infants in Egypt: a quasi-experimental study. Int Breastfeed J. 2008 Nov 21;3:27. doi: 10.1186/1746-4358-3-27. PMID 19025602